CLINICAL TRIAL: NCT05808647
Title: A Randomized Cross-over Study of Low Energy Availability on Pituitary Function in Women
Brief Title: Low Energy Availability and Pituitary Function (LEAP Study)
Acronym: LEAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 22-1811
Record Dates: First submitted 2023-03-29; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Hypogonadotropic Hypogonadism
MeSH Terms: conditions — Hypogonadism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Energy balanced metabolic diet (5-days) (Active Comparator): 45 kcals/kg of fat free mass [FFM]/day; 28% fat, 15% protein, 57% carbohydrate
  Interventions: Behavioral: 5-day controlled metabolic dietary intake
- Low energy availability metabolic diet (5-days) (Experimental): 20 kcal/kg of FFM/day; 28% fat, 15% protein, 57% carbohydrate
  Interventions: Behavioral: 5-day controlled metabolic dietary intake

INTERVENTIONS:
Behavioral: 5-day controlled metabolic dietary intake — Over 5-days, all food will be provided from the metabolic kitchen and participants will be instructed to eat all of the food provided each day and only the food provided each day.

SUMMARY:
The purpose of this study is to learn more about reproductive hormones and if they change in response to 5-days eating an individualized, standardized diet at two levels: energy balance and low energy intake.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18-30
* Body mass index between 18.5-24.9 OR 30-45
* Have regular menstrual cycles between 18-40 days over the past 6 months
* Weight stable (not gained or lost 5kg) in the past 3 months

Exclusion Criteria:

* Using hormonal birth control currently or within the past three months
* Polycystic ovary syndrome (current or past diagnosis)
* Pregnant, lactating, planning to become pregnant in next 6 months
* Engaging in regular intentional aerobic exercise
* Significant medical issues (e.g.,cardiovascular disease or diabetes)

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in stimulated pituitary function, as measured by Luteinizing hormone (LH) area under the curve (AUC) over two hours following pituitary stimulation with a physiologic bolus intravenous dose of gonadorelin acetate | Baseline, ~4-weeks, ~8-weeks (visits timed to to days 1-5 of the menstrual cycle)
  Within-participant changes in response to both conditions will be measured, with lower LH AUC indicating a blunted pituitary response to stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Ann E Caldwell, PhD, Principal Investigator — University of Colorado Anschutz School of Medicine
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months after publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal.